CLINICAL TRIAL: NCT06675149
Title: Effect of Diacutaneus Fibrolysis on Tempromandibular Joint Pain and Trismus Post Oral and Maxillofacial Surgery
Brief Title: Diacutaneus Fibrolysis on Tempromandibular Joint Pain and Trismus Post Oral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aliaa Elsayed Ali, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012/005335
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Massage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (Experimental): This group includes 30 patients who will receive 4 weeks(3times/week) DiacutaneusFibrolysis in addition to post-surgical traditional physiotherapy .
  Interventions: Device: Diacutaneus fibrolysis; Device: Transcutaneous electrical nerve stimulation; Procedure: Massage
- Group A (Placebo Comparator): This group will includes 30 patients who will receive 4 weeks (3times/week) post-surgical traditional physiotherapy (TENS , massage , range of motion exercise ) .
  Interventions: Device: Transcutaneous electrical nerve stimulation; Procedure: Massage

INTERVENTIONS:
Device: Diacutaneus fibrolysis — Material : Stainless steel large angle and small long angle: length 22cm x height 6cm x width 2cm. Weight: 70 grams
  Other Names: Hook measurements
  Arms: Group B
Device: Transcutaneous electrical nerve stimulation — physical therapy electrical modality
  Other Names: TENS
Procedure: Massage — manual therapy intervention

SUMMARY:
This study is carried out on sixty patients who will have tempromandibular pain and trismuspostOral and Maxillofacial Surgeryand their ages will be ranged from 18 to 40 years.

ELIGIBILITY:
Inclusion Criteria:

1. Ages of patients will be ranged from 18 to 40 years.
2. All patients will have Oral and Maxillofacial Surgery.
3. All patients will be referred by a surgeon before starting the study procedure.
4. All participants will have pain and trismus in the jaw,
5. The participants will be also cleared for periodontal issues.
6. All patients will enter the study having their informed consent

Exclusion Criteria:

1. Patients with associated vascular injuries requiring arterial repair.
2. Patient with systemic diseases such as arthritis; pain attributable to confirmed migraine, head, or neck pain condition
3. Patient with acute infection or other significant disease of the teeth, ears, eyes, nose, or throat
4. Patient with present neurologic or cognitive deficit.
5. Patients with history of previously failed surgeries.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
temporomandibular joint pain | pre intervention and re assessed after 1 month
  pain is assessed Pressure pain threshold(PPT) will be obtained with the aid of an algometer by applying pressure to the masseter and to the anterior, middle, and posterior temporalis, increasing pressure until the patient will feel that the pressure will become unpleasant or "painful .
Trismus | pre intervention and re assessed after 1 month
  Trismus is assessed by caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt